CLINICAL TRIAL: NCT05445024
Title: Combination of Nalbuphine and Dexmedetomidine Versus Sufentanil and Dexmedetomidine on Patients After Laparoscopic Gastrointestinal Surgery: A Double-blind, Randomized, Controlled Clinical Study
Brief Title: Combination of Nalbuphine and Dexmedetomidine Versus Sufentanil and Dexmedetomidine on Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LM-WWW-2022
Record Dates: First submitted 2022-04-25; First posted 2022-07-06 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Laparoscopic; Gastrointestinal Surgery
Keywords: laparoscopic; gastrointestinal surgery; nalbuphine; sufentanil; patient-controlled intravenous analgesia; dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nalbuphine group (Experimental): nalbuphine ED95, dexmedetomidine ED95 and ondansetron 16mg were added into normal saline to a total of 100ml
  Interventions: Procedure: nalbuphine group
- sufentanil group (Placebo Comparator): sufentanil (1/1000* nalbuphine ED95), dexmedetomidine ED95 and ondansetron 16mg were added into normal saline to a total of 100ml
  Interventions: Procedure: sufentanil group

INTERVENTIONS:
Procedure: nalbuphine group — nalbuphine ED95, dexmedetomidine ED95 and ondansetron 16mg were added into normal saline to a total of 100ml
  Arms: nalbuphine group
Procedure: sufentanil group — sufentanil (1/1000* nalbuphine ED95), dexmedetomidine ED95 and ondansetron 16mg were added into normal saline to a total of 100ml
  Arms: sufentanil group

SUMMARY:
Surgical pain refers to pain that occurs immediately after surgery, including physical pain and visceral pain. Thus, it severely challenges the proper use of analgesics for patients undergoing laparoscope gastrointestinal surgery to clinicians.

Nalbuphine is a mixed agonist-antagonist opioid. The investigators hypothesized that the clinical effect of nalbuphine in combination with dexmedetomidine might be different from that of sufentanil in combination with dexmedetomidine.

So, the investigators performed a nalbuphine and dexmedetomidine dose finding study, for the patient controlled anaesthesia (PCA) after the laparoscopic gastrointestinal surgery, to establish their 95% effective dose (ED95). The investigators then compared the clinical effect and adverse events of the newly established dosing regimen of nalbuphine combined with dexmedetomidine, to the equivalent dosing of sufentanil combined with dexmedetomidine, in the same patient population.

DETAILED DESCRIPTION:
Surgical pain refers to pain that occurs immediately after surgery, including physical pain and visceral pain. Appropriate perioperative analgesia is a fundamental component of enhanced recovery after surgery. Especially, 45% of postoperative patients experience inadequate pain after gastrointestinal surgery, and uncontrolled postoperative pain prompts respiratory distress, delays wound healing, and a potentially eventual transition from acute to chronic pain problems. Thus, it severely challenges the proper use of analgesics for patients undergoing laparoscope gastrointestinal surgery to clinicians.

Sufentanil is one of the most common opioid used in patient-controlled analgesia (PCA), it may induce many adverse events including respiratory depression, nausea, vomiting, constipation, urinary retention, pruritus, and drowsiness. Many drugs have been combined with dexmedetomidine in PCA to augment analgesic effect or to reduce the adverse events.

Nalbuphine is a mixed agonist-antagonist opioid. Nalbuphine derives its analgesic and sleep-producing effects through agonism at the kappa-opioid receptor with fewer opioid-induced adverse effects. some articles show that it also has the potential to attenuate the mu-opioid receptor-related adverse events. The investigators hypothesized that the clinical effect of nalbuphine in combination with dexmedetomidine might be different from that of sufentanil in combination with dexmedetomidine. Unfortunately, the optimal dosing of nalbuphine combined with dexmedetomidine for the PCIA after the laparoscopic gastrointestinal surgery, has not been determined.

So, the investigators performed a nalbuphine and dexmedetomidine dose finding study, for the PCIA after the laparoscopic gastrointestinal surgery, to establish their 95% effective dose (ED95). The investigators then compared the clinical effect and adverse events of the newly established dosing regimen of nalbuphine combined with dexmedetomidine, to the equivalent dosing of sufentanil combined with dexmedetomidine, in the same patient population.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years and ≤75 years;
2. scheduled to undergo laparoscopic gastrointestinal surgery, under general anaesthesia;
3. 18.5 kg/m2≤BMI≤27.9kg /m2;
4. American Society of Anesthesiology (ASA) I-III;
5. agree to participate, and give signed written informed consents;
6. Verbal or reading ability, able to understand and complete the questionnaire independently or with the help of doctors.

Exclusion Criteria:

1. patients who were allergic to the drugs in this study, who refused to use analgesic devices and analgesic drugs after operation, or who refused to sign the consent forms were not included;
2. severe hypertension, severe psychiatric disease and mental system diseases, severe respiratory diseases, hyperthyroidism, severe liver and kidney dysfunction, alcohol or drug abuse, Severe heart dysfunction or pulmonary insufficiency,Previous history of schizophrenia, epilepsy, myasthenia gravis or delirium;
3. Patients who had a history of drug abuse, patients undergoing chemotherapy and radiotherapy one month before operation, patients unwilling to cooperate with the treatment or with disabilities, were excluded from the study;
4. Patients with a definite diagnosis of chronic pain syndrome, or substance use disorder, patients who used sedatives, antiemetics, or anti-pruritic agents within 24 h before operation;
5. participating in other clinical studies in recent 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) at rest | At 24 hour after operation
  VAS = a 10 cm VAS for pain (0, no pain; 10, worst imaginable pain)

SECONDARY OUTCOMES:
VAS upon movement | Before leaving post anesthesia care(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  VAS = a 10 cm VAS for pain (0, no pain; 10, worst imaginable pain) upon movement (during coughing or changing body position from supine to lateral on bed)
VAS at rest | At 6 hour(T1), 12 hour(T2), 18 hour(T3) ,48 hour(T5) postoperatively.T1 is defined as 6 hour after surgery.T2 is defined as 12 hour after surgery.T3 is defined as 18 hour after surgery.T5 is defined as 48 hour after surgery.
  VAS = a 10 cm VAS for pain (0, no pain; 10, worst imaginable pain)
VAS at rest | Before leaving post anesthesia care unit (PACU)(T0) .T0 is defined as before the patients leave PACU.
  VAS= a 10 cm VAS for pain (0, no pain; 10, worst imaginable pain) at rest
Brinell comfort score (BCS) | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  the Brinell Comfort Score (BCS) 0. for persistent pain;
  1. No pain when quiet, severe pain when deep breathing or coughing;
  2. No pain when quiet, mild pain when deep breathing or coughing;
  3. No pain when quiet and deep breathing;
  4. No pain when coughing.
pressing times of PCIA | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  PCIA(patient controled anesthesia), effective pressing times of PCIA/actual pressing times of PCIA
The number of patients who required remedial analgesic during the first 48h after operation | Within 48hours after surgery
  The number of patients who required remedial analgesic such as opioids(demerol,sufentanil,morphine)or non-steroid anti-inflammatory drugs(acetaminophen,diclofenac).
Frequency of remedial analgesic during the first 48h after operation | Within 48hours after surgery
  Frequency of remedial analgesic during the first 48h after operation
The cumulative remedial analgesic consumption during the first 48h after operation | Within 48hours after surgery
  The cumulative remedial analgesic consumption such as demerol, sufentanil, morphine
PONV | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  PONV (Postoperative nausea and vomiting)=Nausea is defined as subjective,unpleasant sensation associated with awareness of the urge to vomit. Retching is defined as the laboured, spastic, rhythmic contraction of the respiratory muscles without expulsion of the gastric contents.Vomiting is defined as the forceful expulsion of gastric contents from the mouth。0 is no nausea and vomiting; Grade I was nausea without vomiting. Grade Ⅱ was nausea with mild vomiting. Degree III was severe vomiting requiring further treatment. Grade Ⅳ is uncontrollable vomiting.
  The total number of episodes of vomiting was recorded.
pruritus | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  0, no; 1, mild; 2, moderate; 3, severe.
Frequency of remedial antiemetic during the first 48h after operation | Within 48hours after surgery
  Frequency of remedial antiemetic during the first 48h after operation
The cumulative remedial antiemetic consumption during the first 48h after operation | Within 48hours after surgery
  The cumulative remedial antiemetic consumption during the first 48h after operation
Ramsay sedation score | Before leaving PACU(T0) and at 6hour(T1), 12hour(T2), 18hour(T3), 24hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48h postoperatively, respectively.
  Ramsay sedation score (1, anxious, agitated, or restless; 2, cooperative, oriented, and tranquil; 3, responsive to command; 4, briskly responsive; 5, a sluggish response; 6, no response)
The number of patients who required remedial antiemetic during the first 48h after operation | Within 48hours after surgery
  The number of patients who required remedial antiemetic
hypotension | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  Hypotension was defined as systolic arterial pressure <90 mmHg at any investigated time or mean artetial pressure (MAP) decreased by 30% from baseline..
respiratory depression | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  Respiratory depression was defined as ventilatory frequency,8 min-1 or hypoxaemia (SpO2<90%).
dizziness | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  0, no; 1, mild; 2, moderate; 3, severe.
sufentanil | Before leaving PACU(T0). T0 is defined as before the patients leave PACU.
  Sufentanil amount in intraoperative and PACU
Satisfaction rating | T5 is defined as 48 hour after surgery.
  Patients and clinicians were evaluated from three aspects: analgesia effect, sedation and overall evaluation.(0, very dissatisfied;100 points, very satisfied.Score according to actual situation)
HR | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) ad 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48hour postoperatively, respectively.
  heart rate
NBP | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  noninvasive arterial pressure,
SpO2 | Before leaving PACU(T0) and at 6 hour(T1), 12 hour(T2), 18 hour(T3), 24 hour(T4) and 48 hour (T5)postoperatively.T0 is defined as before the patients leave PACU.T1-T5 were defined as 6,12,18,24 and 48 hour postoperatively, respectively.
  oxygen saturation
Time for leaving the bed | at discharge (assessed up to day 7)
  Time for patients to leave the bed and walk
Time for intestinal movement | at discharge (assessed up to day 7)
  Intestinal movement=The patient passed gas for the first time
Time for drinking | at discharge (assessed up to day 7)
  Time for drinking= The patient drink water for the first time
Time for eating | at discharge (assessed up to day 7)
  Time for eating= The patient eat food for the first time

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lv, doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- Meng-Lv, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No